# TaiMed Biologics, Inc.

## Protocol TMB-311 NCT02707861

A Phase 3, Multicenter, Expanded Access Study of Ibalizumab Plus an Optimized Background Regimen (OBR) in Treatment-Experienced Patients Infected With Multi-Drug Resistant (MDR) HIV-1

# Statistical Analysis Plan

August 17, 2018 Final Version 3

TaiMed Biologics, Inc 2 Executive Circle, Suite 280 Irvine, CA 92614

Prepared By: Ken Gerald, PhD Director of Biostatistics

Jennifer Fulton, MS Biostatistician

Westat 5615 Kirby Drive, Suite 710 Houston, TX 77005

**CONFIDENTIAL** 

## **Table of Contents**

| 1. Introduction. 3 2. Study Overview 3 2.1. Study Design 3 2.2. Study Objectives. 4 2.2.1. Primary 4 2.2.2. Secondary 5 2.3. Study Drug Dosage and Administration 5 2.4. Procedures 6 2.4.1. Patient Identification 6 2.4.2. Randomization 6 2.4.3. Blinding/Unblinding 6 2.4.4. Replacement 6 3. Statistical Analysis Considerations 6 3.1. Sample Size 6 3.2. Analysis Populations 6 3.2.1. Intent-to-Treat (ITT) Population 6 3.2.2. Safety (SAF) Population 7 3.3. Data Handling 7 3.3.1. Measurement Times 7 3.3.2. Clinical Laboratory Data Handling Conventions 7 3.3.3. Baseline Values 7 3.3.4. Missing Data Conventions 8 3.4. Statistical Methods 8 3.4.1. General Overview and Plan of Analysis 8 3.4.1. General Overview and Plan of Analysis 9 4. Statistical Analysis 9 |
|---|
| 2.1. Study Objectives. 3 2.2. Study Objectives. 4 2.2.1. Primary. 4 2.2.2. Secondary. 5 2.3. Study Drug Dosage and Administration 5 2.4. Procedures. 6 2.4.1. Patient Identification 6 2.4.2. Randomization 6 2.4.3. Blinding/Unblinding. 6 2.4.4. Replacement 6 3. Statistical Analysis Considerations. 6 3.1. Sample Size 6 3.2. Analysis Populations. 6 3.2.1. Intent-to-Treat (ITT) Population 6 3.2.2. Safety (SAF) Population 7 3.3. Data Handling. 7 3.3.1. Measurement Times 7 3.3.2. Clinical Laboratory Data Handling Conventions 7 3.3.3. Baseline Values 7 3.3.4. Missing Data Conventions 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Clinical Laboratory Para |
| 2.1. Study Objectives. 3 2.2. Study Objectives. 4 2.2.1. Primary. 4 2.2.2. Secondary. 5 2.3. Study Drug Dosage and Administration 5 2.4. Procedures. 6 2.4.1. Patient Identification 6 2.4.2. Randomization 6 2.4.3. Blinding/Unblinding 6 2.4.4. Replacement 6 3. Statistical Analysis Considerations 6 3.1. Sample Size 6 3.2. Analysis Populations 6 3.2.1. Intent-to-Treat (ITT) Population 6 3.2.2. Safety (SAF) Population 7 3.3. Data Handling 7 3.3.1. Measurement Times 7 3.3.2. Clinical Laboratory Data Handling Conventions 7 3.3.3. Baseline Values 7 3.3.4. Missing Data Conventions 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Clinical Laboratory Paramete |
| 2.2. Study Objectives 4 2.2.1. Primary 4 2.2.2. Secondary 5 2.3. Study Drug Dosage and Administration 5 2.4. Procedures 6 2.4.1. Patient Identification 6 2.4.2. Randomization 6 2.4.3. Blinding/Unblinding 6 2.4.4. Replacement 6 3. Statistical Analysis Considerations 6 3.1. Sample Size 6 3.2. Analysis Populations 6 3.2.1. Intent-to-Treat (ITT) Population 6 3.2.2. Safety (SAF) Population 7 3.3.1. Measurement Times 7 3.3.2. Clinical Laboratory Data Handling Conventions 7 3.3.3. Baseline Values 7 3.3.4. Missing Data Conventions 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.2. AEs 10 4.3.3. Clinical Laborator |
| 2.2.2. Secondary. 5 2.3. Study Drug Dosage and Administration 5 2.4. Procedures. 6 2.4.1. Patient Identification 6 2.4.2. Randomization 6 2.4.3. Blinding/Unblinding. 6 2.4.4. Replacement 6 3. Statistical Analysis Considerations 6 3.1. Sample Size. 6 3.2. Analysis Populations. 6 3.2.1. Intent-to-Treat (ITT) Population 6 3.2.2. Safety (SAF) Population 7 3.3. Data Handling. 7 3.3.1. Measurement Times 7 3.3.2. Clinical Laboratory Data Handling Conventions 7 3.3.3. Baseline Values. 7 3.3.4. Missing Data Conventions 8 3.4. Statistical Methods. 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Clinical Laboratory Parameters 10 4.3.2. AEs 10 4.3.4. Vital Si |
| 2.2.2. Secondary. 5 2.3. Study Drug Dosage and Administration 5 2.4. Procedures. 6 2.4.1. Patient Identification 6 2.4.2. Randomization 6 2.4.3. Blinding/Unblinding. 6 2.4.4. Replacement 6 3. Statistical Analysis Considerations 6 3.1. Sample Size. 6 3.2. Analysis Populations. 6 3.2.1. Intent-to-Treat (ITT) Population 6 3.2.2. Safety (SAF) Population 7 3.3. Data Handling. 7 3.3.1. Measurement Times 7 3.3.2. Clinical Laboratory Data Handling Conventions 7 3.3.3. Baseline Values. 7 3.3.4. Missing Data Conventions 8 3.4. Statistical Methods. 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Clinical Laboratory Parameters 10 4.3.2. AEs 10 4.3.4. Vital Si |
| 2.3. Study Drug Dosage and Administration 5 2.4. Procedures 6 2.4.1. Patient Identification 6 2.4.2. Randomization 6 2.4.3. Blinding/Unblinding 6 2.4.4. Replacement 6 3. Statistical Analysis Considerations 6 3.1. Sample Size 6 3.2. Analysis Populations 6 3.2.1. Intent-to-Treat (ITT) Population 6 3.2.2. Safety (SAF) Population 7 3.3. Data Handling 7 3.3.1. Measurement Times 7 3.3.2. Clinical Laboratory Data Handling Conventions 7 3.3.3. Baseline Values 7 3.3.4. Missing Data Conventions 8 3.4. Statistical Methods 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 12 |
| 2.4.1. Patient Identification 6 2.4.2. Randomization 6 2.4.3. Blinding/Unblinding 6 2.4.4. Replacement 6 3. Statistical Analysis Considerations 6 3.1. Sample Size 6 3.2. Analysis Populations 6 3.2.1. Intent-to-Treat (ITT) Population 6 3.2.2. Safety (SAF) Population 7 3.3. Data Handling 7 3.3.1. Measurement Times 7 3.3.2. Clinical Laboratory Data Handling Conventions 7 3.3.3. Baseline Values 7 3.3.4. Missing Data Conventions 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 2.4.2. Randomization 6 2.4.3. Blinding/Unblinding 6 2.4.4. Replacement 6 3. Statistical Analysis Considerations 6 3.1. Sample Size 6 3.2. Analysis Populations 6 3.2.1. Intent-to-Treat (ITT) Population 6 3.2.2. Safety (SAF) Population 7 3.3. Data Handling 7 3.3.1. Measurement Times 7 3.3.2. Clinical Laboratory Data Handling Conventions 7 3.3.3. Baseline Values 7 3.3.4. Missing Data Conventions 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.5. Physical Examination Findings 12 |
| 2.4.3. Blinding/Unblinding 6 2.4.4. Replacement 6 3. Statistical Analysis Considerations 6 3.1. Sample Size 6 3.2. Analysis Populations 6 3.2.1. Intent-to-Treat (ITT) Population 6 3.2.2. Safety (SAF) Population 7 3.3. Data Handling 7 3.3.1. Measurement Times 7 3.3.2. Clinical Laboratory Data Handling Conventions 7 3.3.3. Baseline Values 7 3.3.4. Missing Data Conventions 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 2.4.4. Replacement 6 3. Statistical Analysis Considerations 6 3.1. Sample Size 6 3.2. Analysis Populations 6 3.2.1. Intent-to-Treat (ITT) Population 6 3.2.2. Safety (SAF) Population 7 3.3.1. Measurement Times 7 3.3.2. Clinical Laboratory Data Handling Conventions 7 3.3.3. Baseline Values 7 3.3.4. Missing Data Conventions 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 2.4.4. Replacement 6 3. Statistical Analysis Considerations 6 3.1. Sample Size 6 3.2. Analysis Populations 6 3.2.1. Intent-to-Treat (ITT) Population 6 3.2.2. Safety (SAF) Population 7 3.3.1. Measurement Times 7 3.3.2. Clinical Laboratory Data Handling Conventions 7 3.3.3. Baseline Values 7 3.3.4. Missing Data Conventions 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 3.1. Sample Size 6 3.2. Analysis Populations 6 3.2.1. Intent-to-Treat (ITT) Population 6 3.2.2. Safety (SAF) Population 7 3.3. Data Handling 7 3.3.1. Measurement Times 7 3.3.2. Clinical Laboratory Data Handling Conventions 7 3.3.3. Baseline Values 7 3.3.4. Missing Data Conventions 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 3.2. Analysis Populations 6 3.2.1. Intent-to-Treat (ITT) Population 6 3.2.2. Safety (SAF) Population 7 3.3. Data Handling 7 3.3.1. Measurement Times 7 3.3.2. Clinical Laboratory Data Handling Conventions 7 3.3.3. Baseline Values 7 3.3.4. Missing Data Conventions 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 3.2. Analysis Populations 6 3.2.1. Intent-to-Treat (ITT) Population 6 3.2.2. Safety (SAF) Population 7 3.3. Data Handling 7 3.3.1. Measurement Times 7 3.3.2. Clinical Laboratory Data Handling Conventions 7 3.3.3. Baseline Values 7 3.3.4. Missing Data Conventions 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 3.2.2. Safety (SAF) Population 7 3.3. Data Handling 7 3.3.1. Measurement Times 7 3.3.2. Clinical Laboratory Data Handling Conventions 7 3.3.3. Baseline Values 7 3.3.4. Missing Data Conventions 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 3.2.2. Safety (SAF) Population 7 3.3. Data Handling 7 3.3.1. Measurement Times 7 3.3.2. Clinical Laboratory Data Handling Conventions 7 3.3.3. Baseline Values 7 3.3.4. Missing Data Conventions 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 3.3. Data Handling |
| 3.3.1. Measurement Times 7 3.3.2. Clinical Laboratory Data Handling Conventions 7 3.3.3. Baseline Values 7 3.3.4. Missing Data Conventions 8 3.4. Statistical Methods 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 3.3.3. Baseline Values 7 3.3.4. Missing Data Conventions 8 3.4. Statistical Methods 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 3.3.3. Baseline Values 7 3.3.4. Missing Data Conventions 8 3.4. Statistical Methods 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 3.3.4. Missing Data Conventions 8 3.4. Statistical Methods 8 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 3.4.1. General Overview and Plan of Analysis 8 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 3.4.2. Hypothesis Testing 9 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 4. Statistical Analysis 9 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 4.1. Patient Disposition 9 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 4.2. Demographic and Physical Characteristics 9 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 4.3. Analysis of Safety and Tolerability 10 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 4.3.1. Extent of Study Drug Exposure 10 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 4.3.2. AEs 10 4.3.3. Clinical Laboratory Parameters 11 4.3.4. Vital Signs 12 4.3.5. Physical Examination Findings 12 |
| 4.3.4. Vital Signs |
| 4.3.5. Physical Examination Findings |
| and the second of the second o |
| 4.3.6. Medications |
| 4.4. Efficacy |
| 4.5.1. Primary Efficacy Endpoint |
| 4.5.2. Secondary Efficacy Endpoints |
| 4.5.3. Graphical Displays |
| 4.6. Exploratory/Other Analyses |
| 5. References |
| 6. Proposed Summary Listings and Tables |

#### 1. Introduction

This document outlines the planned statistical analyses for data collected within the scope of the TaiMed ibalizumab protocol TMB-311, entitled "A Phase 3, Multicenter, Expanded Access Study of Ibalizumab Plus an Optimized Background Regimen (OBR) in Treatment-Experienced Patients Infected With Multi-Drug Resistant (MDR) HIV-1". This statistical analysis plan (SAP) applies to the most recent version of the study protocol (dated 11 December 2017) and will be updated as necessary if future protocol amendments warrant an update to the manner of analysis. This document was prepared in accordance with the International Conference on Harmonisation (ICH) Guideline E3: Structure and Content of Clinical Study Reports [1].

#### 2. Study Overview

#### 2.1. Study Design

This Phase 3 multicenter study will evaluate safety and tolerability of ibalizumab in HIV positive patients with MDR HIV infection. Eligible patients will include those currently receiving ibalizumab under a TaiMed-sponsored or Investigator-INDprotocol, and treatment-experienced patients with no history of ibalizumab treatment who are on a failing regimen, or who have failed and are off treatment. Patients will be enrolled in one of two Cohorts. Cohort 1 consists of patients currently receiving ibalizumab via other TaiMed-sponsored or Investigator-IND (compassionate use) protocols. These patients will continue their current dosage of ibalizumab (800 mg every 2 weeks or 2000 mg every 4 weeks). Cohort 2 consists of patients initiating ibalizumab. These patients will receive a 2000 mg loading dose at Baseline/Day 0 followed by 800 mg maintenance doses every 2 weeks.

For Cohort 1, screening procedures and Day 0 procedures are scheduled for the same day. Patients who qualify for entry into Cohort 1 of this study who are currently receiving 800 mg ibalizumab every 2 weeks will have physical and laboratory measures performed and receive the first on-study dose of ibalizumab at Screening/Day 0. These patients will return to the clinic on Day 14 and every 2 weeks thereafter through the remainder of participation in the study (up to 144 weeks) for study drug administration (800 mg) and effectiveness and safety evaluations. Patients who are discontinued or who withdraw from the study prematurely will be asked to return for an Early Withdrawal visit to have all assessments detailed in the Schedule of Events for that visit performed.

Patients who qualify for entry into Cohort 1 of this study who are currently receiving 2000 mg ibalizumab every 4 weeks will have physical and laboratory measures performed, and receive the first on-study dose of ibalizumab at Screening/Day 0. These patients will return to the clinic at Week 4 and every 4 weeks thereafter through the remainder of participation in the study (up to 144 weeks) for study drug administration (2000 mg) and effectiveness and safety evaluations. Patients who are discontinued or who withdraw from the study prematurely will be asked to return for

an Early Withdrawal visit to have all assessments detailed in the Schedule of Events for that visit performed.

For Cohort 2, patients will complete all screening procedures during the six weeks before Baseline/Day 0. Successful screening results will allow the patients to proceed to the Baseline/ Day 0 Visit, where they will initiate the selected OBR in addition to undergoing physical and laboratory measures. At this visit patients will also receive the loading dose of the study medication (2000 mg). Patients will return to the clinic on Day 7 for effectiveness and safety evaluations, and on Day 14 and every two weeks thereafter through the remainder of participation in the study (up to 144 weeks) for study drug administration (800 mg) and effectiveness and safety evaluations. Patients who are discontinued or who withdraw from the study prematurely will be asked to return for an Early Withdrawal visit to have all assessments detailed in the Schedule of Events for that visit performed.

All patients who complete Week 144 or end of study (EOS) visit will return for a follow-up visit at Week 150. Patients may be discontinued from the study at the patient's request or if the patient becomes pregnant, at investigator request, for a protocol violation, for treatment-related serious or intolerable adverse events (AEs), for toxicity (defined as two consecutive laboratory results, at least 14 days apart, with a CD4+ T-cell count below 200 cells/mm3 that also represents a 50% reduction from the Baseline CD4+ T-cell count), or for virologic failure. Virologic failure is defined as two consecutive measurements beginning at Week 24 or later if less than a 0.5 log10 decline from the Baseline viral load.

## 2.2. Study Objectives

## 2.2.1. Primary

The primary objectives of this study are to:

#### Cohort 1

- Continue to provide ibalizumab to patients currently receiving ibalizumab treatment under Investigator-sponsored INDs or TaiMed-sponsored protocols
- Demonstrate the safety and tolerability of ibalizumab in HIV positive patients with MDR HIV infection

#### Cohort 2

- Provide access to ibalizumab for qualifying MDR HIV-1 infected patients with limited treatment options
- Demonstrate the safety, efficacy, and tolerability of ibalizumab in HIV positive patients with MDR HIV infection

## 2.2.2. Secondary

The secondary objectives of this study are to:

- Demonstrate the antiviral activity of ibalizumab in HIV positive patients with MDR HIV infection
- Characterize HIV-1 sensitivity/susceptibility changes associated with protocol-defined virologic failure after ibalizumab administration in combination with OBR
- Determine the presence and significance of anti-ibalizumab antibodies associated with protocol-defined virologic failure after ibalizumab administration, if any (immunogenicity of ibalizumab)

#### 2.3. Study Drug Dosage and Administration

The investigational product, ibalizumab, is a humanized IgG4 monoclonal antibody (MAb) administered via intravenous (IV) infusion. Patients will be enrolled in one of two Cohorts (Cohort 1 and Cohort 2). Cohort 1 patients will continue their current dosage of ibalizumab (800 mg every 2 weeks or 2000 mg every 4 weeks). Cohort 2 patients will receive a 2000 mg loading dose at Baseline/Day 0 followed by 800 mg maintenance doses every 2 weeks.

Patients receiving ibalizumab under Investigator-IND protocols, who will enroll into Cohort 1 of this study, are currently being supplied with ibalizumab vials containing a 1.2 mL injection volume and 180 mg ibalizumab per vial. For this study, these patients will continue receiving ibalizumab in this vial configuration until that supply of drug product is exhausted, at which time they will be switched to the drug product with a 1.33 mL injection volume and 200 mg ibalizumab per vial.

Patients receiving ibalizumab in study TMB-301, who will enroll into Cohort 1 of this study, and patients initiating ibalizumab in Cohort 2 will receive only vials with a 1.33 mL injection volume and 200 mg ibalizumab per vial. During this study, it will be very important to ensure that all drug supplies are clearly labeled and segregated by vial configuration to prevent confusion.

In addition to the study drug, all patients will receive an OBR, which is a standard—of-care regimen selected by the investigator based upon treatment history and the results of recent viral resistance testing. For patients enrolling into Cohort 2, previous resistance testing done within 6 months prior to Screening must demonstrate that the patient's viral isolate is sensitive/susceptible to a minimum of one of the agents selected for the OBR. The patient must be willing and able to take at least one of the agents to which their virus is sensitive/susceptible as part of the OBR.

#### 2.4. Procedures

#### 2.4.1. Patient Identification

Once consent is obtained and study eligibility has been determined, a patient will be enrolled into the study and will be assigned a Participant Identification (PID) number. The 5-digit PID number will consist of a 2-digit site number and a 3-digit sequential patient number. If a patient in Cohort 2 is a screen failure, the PID number will not be reassigned.

## 2.4.2. Randomization

This will be an open-label, non-randomized study.

## 2.4.3. Blinding/Unblinding

There will be no blinding/unblinding considerations for this open-label, non-randomized study.

## 2.4.4. Replacement

Patients who withdraw or otherwise discontinue the study prematurely will not be replaced.

## 3. Statistical Analysis Considerations

#### 3.1. Sample Size

Anticipated enrollment is approximately 100 patients from approximately 50 sites in North America; however, the numbers of participating patients and sites will not be limited and may exceed 100 patients.

## 3.2. Analysis Populations

## 3.2.1. Intent-to-Treat (ITT) Population

The ITT population is defined as all patients enrolled into the TMB-311 study. The ITT Analysis Population will be used for the patient disposition, demographic and physical characteristics, and efficacy analyses.

If there are ITT patients who do not receive at least one complete dose of study drug, then a modified ITT (mITT) Analysis Population will be used for a supportive effectiveness analysis.

## 3.2.2. Safety (SAF) Population

All patients who receive at least one partial dose of study drug will be included in the SAF Population. Patients will be analyzed according to the treatment they actually received. The SAF Population will be used for the safety analyses.

#### 3.3. Data Handling

#### 3.3.1. Measurement Times

The nominal visit time point entered on the electronic case report forms (eCRFs) will be used. Patients are asked to adhere to the following visit schedule (with windows in parentheses):

- For Cohort 1 patients, Screening and Day 0 (first on-study administration of ibalizumab) are scheduled for the same day.
- For Cohort 2 patients, the Screening will occur 1 to 6 weeks prior to Day 0.
- For Cohort 2, Day 7 (+/- 1 day) serves as the time point at which the antiviral activity of ibalizumab will be assessed to address the primary effectiveness objective.
- For all Cohorts, Day 14 (+/- 1 day) and Week 4 (+/- 2 days) through Week 144/EOS Visit (+/- 2 days) from the Day 0 date (Visit Week will depend on the dosing schedule per Cohort 1 or 2; please refer to the Schedule of Visits Tables 3.1-3.6 in the study protocol).

## 3.3.2. Clinical Laboratory Data Handling Conventions

If a patient has multiple results in the clinical laboratory data for the Screening visit, only the last result prior to the first dose of study drug will be included in the analysis. If a patient has multiple results (retests) for subsequent visits, the retest results will only be included in the analysis if the patient does not have a value recorded for the original assessment at the given visit.

#### 3.3.3. Baseline Values

For patients in Cohort 1 who were enrolled in the TMB-202 or TMB-301 studies, Baseline values for TMB-311 are defined as the values recorded for the Baseline visit in the previous study. For patients in Cohort 1 who were not enrolled in the TMB-202 or TMB-301 studies as well as for patients in Cohort 2, Baseline is defined as the last assessment prior to their first dose of study drug on the TMB-311 Day 0 visit.

## 3.3.4. Missing Data Conventions

Cohort 2 patients with missing data at Day 0 will use the Screening visit value as their Day 0 result. Similarly, patients with missing data at Screening will use the Day 0 visit value as their Screening result. No Screening or Day 0 data will be imputed for Cohort 1 patients.

Unless otherwise specified, missing data for subsequent visits will be considered missing at random and will not be imputed. If necessary, imputation of partial dates may be performed during the data analysis and will be documented (e.g., missing month=July; missing day=15).

The **Missing Equals Failure (MEF)** imputation technique will be applied to the viral load measures (log<sub>10</sub> copies/mL and copies/mL) only. If a viral load measurement is missing at any scheduled visit, the value will be replaced with the baseline viral load measurement. Also, all visits after a confirmed virologic failure will be imputed as failures (replaced with the baseline measurement) for all study visits even if the patient discontinued early.

The Last Observation Carried Forward (LOCF) imputation technique will be applied to the CD4+ T-Cell Counts (cells/mm³) only. If a CD4+ T-Cell Count is missing at any scheduled visit, the value will be replaced with the most recent previous non-missing value.

#### 3.4. Statistical Methods

#### 3.4.1. General Overview and Plan of Analysis

The data collected are intended primarily for clinical review and interpretation. The analysis of study data will be primarily descriptive, with emphasis on tabular and graphical displays. Descriptive statistics will be used to guide decisions as to the clinical relevance of findings. Unless otherwise stated, p-values will be determined only if they appear to be warranted from the summary statistics.

All results will be displayed in the following patient groupings:

- 1) Cohort 1 TMB-301 rollover patients;
- 2) Cohort 1 TMB-202 rollover patients in the 800mg dose group;
- 3) Cohort 1 TMB-202 rollover patients in the 2000mg dose group;
- 4) Cohort 2 patients;
- 5) Total includes all patients from 1-4.

The two patients who were formerly enrolled in the investigator-sponsored IND (compassionate use) studies will be included in listings only.

For continuous data, descriptive statistics will be presented as number of patients (n), mean, standard deviation, median, minimum and maximum. For categorical data, the frequency and percentage of patients in each category will be presented. Percentages will be based on non-missing data unless otherwise specified.

Data will be described and analyzed using the SAS System Version 9 (SAS Institute Inc., Cary, NC, SAS System). Individual patient data will be presented in patient data listings.

## 3.4.2. Hypothesis Testing

This study is designed to evaluate the safety and efficacy of ibalizumab in treatment-experienced patients infected with multi-drug resistant HIV-1. No formal statistical hypothesis testing is planned for the study. [Note: Hypothesis testing may be performed as additional/exploratory analyses (see Section 4.6)].

## 4. Statistical Analysis

## 4.1. Patient Disposition

The number of patients in the ITT and SAF Populations will be tabulated.

Study completion data will be summarized for all enrolled patients. The number and percent of patients who complete treatment; discontinue study medication prematurely; or discontinue the study prematurely will be tabulated. The primary reason for premature discontinuation of study medication and/or discontinuation from study participation will be tabulated. Any additional reason(s) for premature discontinuation of study medication will also be tabulated. A listing of all enrolled patients will be provided.

#### 4.2. Demographic and Physical Characteristics

Summary statistics will be presented for demographic and other Baseline characteristics for the ITT Population. Tabulations for age, sex, ethnicity (Hispanic/Latino, Neither Hispanic nor Latino, Unknown), and race (American Indian/Alaska Native, Asian, Black/African American, Native Hawaiian/Other Pacific Islander, White, Unknown, or Other) will be presented. Age (years) will be calculated as the integer part of [(date of screening - date of birth + 1)/365.25]. Baseline physical characteristics, such as height (cm) and weight (kg), will also be summarized.

A listing of demographic and Baseline characteristics will be presented, as well as a listing of medical history.

#### 4.3. Analysis of Safety and Tolerability

Safety and tolerability will be assessed by both clinical and laboratory examinations. Summary statistics will be presented by AEs; hematology and chemistry; vital signs, changes from Baseline, and clinically significant findings; and abnormal physical examination findings in the SAF Population. Clinical laboratory values outside the normal ranges will be flagged in patient data listings. Non-numeric data will be presented in patient data listings, but will not be tabulated.

## 4.3.1. Extent of Study Drug Exposure

Summary statistics will be presented for the cumulative dose (mg) and duration of treatment received by the patients in the SAF Population. Duration of treatment will be represented as number of days from first dose of study drug. For Cohort 1 patients, the date of their first dose of study drug in the previous study will be used. Corresponding listings will also be generated for study drug administration and OBR adherence.

#### 4.3.2. **AEs**

All AEs will be coded, using MedDRA dictionary version 17.0. The use of another version will not be considered a violation of the SAP, nor require an amendment to the plan. All summary tables will be based on coded preferred terms (PTs), instead of verbatim terms. The only exception being all rashes are combined into one category named RASHES. The categories and definitions of severity and causal relationship for all AEs, including the criteria for which an AE is to be classified as "serious," are as described in the protocol (Section 8).

A treatment-emergent AE (TEAE) is defined as any event not present before exposure to study drug or any event already present that worsens in either intensity or frequency following exposure to study drug. AEs with missing start dates, but with stop dates either overlapping into the dosing period or missing, will be considered TEAEs. A TEAE with missing severity or relationship will be considered severe or related, respectively.

The overall incidence of TEAEs will be summarized for all patients in the SAF Population. The number and percentage of patients having the following will be tabulated:

- TEAE
- Serious TEAE
- TEAE leading to discontinuation
- TEAE with outcome of death
- TEAE related to study drug (definitely, probably, or possibly)

- Severe TEAE
- Class C TEAE per the Centers for Disease Control and Prevention (CDC) Classification System for HIV Infection

The overall incidence of TEAEs will also be summarized by System Organ Class (SOC), and by SOC and PT. The number and percentage of patients reporting an event, as well as the number of events reported by the patients will be tabulated. The incidence of serious TEAEs and TEAEs leading to study discontinuation (if any) will be summarized in the same manner. If there are multiple occurrences of the same TEAE within any SOC or PT for the same patient, only the first occurrence will be counted.

The incidence of TEAEs by severity/grade (mild, moderate, severe, or potentially life-threatening) and by relationship to study drug (unrelated, possibly related, probably related, and definitely related), and the incidence of SAEs by relationship to study drug, will also be summarized.

All other AEs will be classified as non-TEAEs and identified in listings only. Serious TEAEs, TEAEs leading to study discontinuation, and TEAEs with an outcome of death will be presented in separate listings, if needed.

These tables will be repeated for patients receiving an investigational agent [Fostemsavir (BMS-068), Cabotegravir, or PRO140] as a concomitant medication versus those patients who did not receive an investigational agent.

#### 4.3.3. Clinical Laboratory Parameters

Summary statistics will be presented for laboratory measurements (hematology and chemistry) overall for all patients in the SAF Population. Urinalysis results will be presented in a listing. The following analytes will be tabulated/listed:

- **Hematology**: complete white blood cell count with differential, hemoglobin, hematocrit, and platelets.
- **Serum chemistry profile**: albumin, alkaline phosphatase, alanine aminotransferase (ALT), amylase, aspartate aminotransferase (AST), blood urea nitrogen, calcium, chloride, creatine phosphokinase, creatinine, direct bilirubin, gamma glutamyl transferase, glucose, lactate dehydrogenase, lipase, lipid profile (total cholesterol, highdensity lipoprotein, low-density lipoprotein, and triglycerides), magnesium, phosphorus, potassium, sodium, total bilirubin, total protein, and uric acid. In addition, eGFR will be presented using the following formula: eGFR = 1.86 x [Creatinine/88.4]<sup>-1.154</sup> x [Age]<sup>-0.203</sup> x [0.742 if female] x [1.210 if Black].

Urinalysis results will be presented in a data listing and will include results from microscopic testing only. Pregnancy test, Serum Follicle-Stimulating Hormone (FSH) test, Hepatitis Serology, C-reactive Protein, and Viral Resistance Testing will also be presented in a data listing only.

Normal ranges for the laboratory parameters will be provided by the laboratory that performed the assessments. All normal ranges will be standardized and results will be reported in standard units. The tables will include summary statistics for the Baseline assessments and the changes from Baseline to each subsequent time point of measurement. A listing of patients with abnormal (i.e., outside normal range) laboratory assessments will also be presented.

Potentially Clinically Significant (PCS) criteria may be applied to laboratory parameters as clinically indicated, and if applied, will be summarized as described above. PCS is defined as a laboratory value that is lower or higher than a laboratory's normal range limits.

Note: Electronic clinical laboratory data will be received at Westat. Data reconciliation will be performed to resolve any discrepancies with the Oracle database. Details of data receipt will be described in the Data Receipt Plan.

## 4.3.4. Vital Signs

Summary statistics for vital signs and weight will be presented overall for all patients in the SAF Population for all scheduled visits. Actual values and changes from Baseline will be summarized for all visits where collected.

## 4.3.5. Physical Examination Findings

Physical examination findings at each scheduled visit will be summarized overall for all patients in the SAF Population. The number and percent of patients with abnormal findings by body system will be tabulated.

## 4.3.6. Medications

All prescriptions or over-the-counter medications continued at the start of the trial or started during the trial, and different from the study drug will be recorded. All of these medications will be coded, using WHO Drug Dictionary (March 2014). The use of another version will not be considered a violation of the SAP, nor require an amendment to the plan. Both the coded terms and verbatim terms will be presented in data listings for:

• Concomitant procedures (procedures are not coded)

- Previous and Concomitant medications
- OBR medications
- ART medications

## 4.4. Efficacy

As described in section 3.3.3 of this document, the MEF technique will be applied to the efficacy analyses with regard to imputing missing viral load results as applicable. Note: Prior to calculating change from Baseline in viral load, the log10 value of each measurement will be calculated and will be rounded to one decimal point.

## 4.5.1. Primary Efficacy Endpoint

Per the protocol, the primary efficacy endpoint for the Cohort 2 patients is defined as the proportion of patients achieving  $a \ge 0.5 \log_{10}$  decrease in viral load from Baseline at Day 7 on study drug. A 95% confidence interval around the observed rate will be presented. This endpoint will be presented for all Cohort 2 patients, as well as stratified by:

- 1) Sex (Male vs Female)
- 2) Age (<50 vs > 50)
- 3) Race (Caucasian, Asian, and Other)

The primary efficacy endpoint will not be analyzed for the TMB-301 and TMB-202 rollover patients, as they did not have dosing or viral load measurements at Day 7 on study drug in the TMB-311 study.

## 4.5.2. Secondary Efficacy Endpoints

Although the TMB-311 protocol indicates the secondary efficacy endpoints would only be performed for the Cohort 2 patients, for completeness all secondary efficacy endpoints will be assessed for all patients in all cohorts at applicable visits.

#### 4.5.2.1 HIV-1 RNA levels (copies/mL)

The frequency and proportion of patients achieving RNA levels < 50 copies/mL and < 400 copies/mL along with 95% confidence intervals around the observed rate will be presented at all key visits [Day 7 (Cohort 2 only), and Weeks 24, 48, 72, 96, 120, and 144/EOS] where assessed.

Summary statistics for the actual and change from Baseline of RNA levels will be presented for at all visits where assessed.

#### 4.5.2.2 Viral Load (log<sub>10</sub> copies/mL)

The frequency and proportion of patients achieving a  $\geq 0.5 \log_{10}$  and  $\geq 1.0 \log_{10}$  decrease from Baseline in viral load along with 95% confidence intervals will be performed at all key visits [Day 7 (Cohort 2 only), and Weeks 24, 48, 72, 96, 120, and 144/EOS] where assessed. The mean change from Baseline at all assessment time points will be presented.

These tables will be repeated for patients receiving an investigational agent [Fostemsavir (BMS-068), Cabotegravir, or PRO140] as a concomitant medication versus those patients who did not receive an investigational agent.

#### 4.5.2.3 Virologic Outcome

## Snapshot Approach

Virologic outcome will be assigned for each patient at each key visit after Week 12 [Weeks 24, 48, 72, 96, 120, and 144/EOS], per the snapshot approach, using the following standard categories:

- 1=Virologic success (≥0.5 log10 decline from Baseline in viral load)
- 2a=(<0.5 log<sub>10</sub> copies/mL drop from Baseline in viral load)
- 2b=Discontinued efficacy portion of study because of virologic failure (may still continue safety)
- 2c=Discontinued because of other reasons and the drop from baseline in viral load at the time of discontinuation was <0.5 log<sub>10</sub> copies/mL
- 2d=OBR changed
- 3a=Discontinued because of AE or death
- 3b=Discontinued because of other reasons and the drop from baseline in viral load at the time of discontinuation was >=0.5 log<sub>10</sub> copies/mL
- 3c=Missing data during the window but on study

## Other Virologic Outcomes

Other virologic outcomes will also be defined as follows:

#### Failure to achieve/maintain response:

Patient does not have  $\ge 0.5 \log_{10}$  decline from baseline (BL) by Week 12 on study drug OR patient has a  $0.5 \log_{10}$  decline from BL prior to Week 12 but fails to maintain the  $0.5 \log_{10}$  decline from BL and does not have a  $\ge 1 \log_{10}$  increase from nadir on any two consecutive scheduled efficacy assessments after achieving the  $\ge 0.5 \log_{10}$  decline from BL.

#### Rebound:

Patient has a  $\ge 0.5 \log 10$  decline from BL by Week 12 but viral load remains  $\ge 50$  copies (not suppressed), followed by  $\ge 1 \log_{10}$  increase from nadir at two consecutive scheduled visits any time after achieving the  $\ge 0.5 \log_{10}$  decline from BL.

#### **Breakthrough:**

Patient has suppressed viral load (< 50 copies) at any time after primary endpoint followed by ≥200 copies at two consecutive scheduled efficacy assessments.

## **Suboptimal Response:**

Patient has a  $\ge 0.5 \log_{10}$  decline but does not suppress (< 50 copies) at any time after primary endpoint and does not have a  $\ge 1 \log_{10}$  increase from nadir on any two consecutive scheduled efficacy assessments after achieving the  $\ge 0.5 \log_{10}$  decline from BL.

## **Virologic Suppression:**

Patient has a  $\ge 0.5 \log_{10}$  decline and does suppress (< 50 copies) at any time after primary endpoint and does not have a  $\ge 1 \log_{10}$  increase from nadir on any two consecutive scheduled efficacy assessments after achieving the  $\ge 0.5 \log_{10}$  decline from BL.

A table summarizing virologic outcome at the each key visit after Week 12 [Weeks 24, 48, 72, 96, 120, and 144/EOS] according to the above categories will be provided. A listing indicating the virologic outcome for each patient will be included.

#### 4.5.2.4 CD4+ T-Cell Counts

Summary statistics will be presented for CD4+ T-cell count and change from Baseline in CD4+ T-cell count at the each key visit after Week 12 [Weeks 24, 48, 72, 96, 120, and 144/EOS].

CD4+ T-Cell Counts for all patients at all assessed visits will also be presented in a data listing. The listing will include a column indicating whether or not the patient met the definition of toxicity (2 consecutive laboratory results, at least 14 days apart, with a CD4+ T-cell count below

200 cells/mm<sup>3</sup> that also represents a 50% reduction from the Baseline CD4+ T-cell count).

## 4.5.3. Graphical Displays

In addition to the tables and listings described above, the following graphical displays of efficacy endpoints will also be included:

- Proportion of patients achieving a ≥ 0.5 log<sub>10</sub> decrease from Baseline in viral load at all scheduled visits;
- Proportion of patients achieving  $a \ge 1.0 \log_{10}$  decrease from Baseline in viral load at all scheduled visits;
- Proportion of patients achieving RNA levels < 50 copies/mL at all scheduled visits;
- Proportion of patients achieving RNA levels < 400 copies/mL at each study visit;
- Mean (+/- SE) RNA levels (copies/mL) at all scheduled visits;
- Mean (+/- SE) change from Baseline in RNA levels (copies/mL) at all scheduled visits;
- Mean (+/- SE) CD4+ cell count (cells/mm<sup>3</sup>) at all scheduled visits;
- Mean (+/- SE) change from Baseline in CD4+ T-cell count (cells/mm<sup>3</sup>) at all scheduled visits.

## 4.6. Exploratory/Other Analyses

Summaries of viral resistance test results, immunogenicity results, and other virology results will be presented, prepared by TaiMed.

#### 5. References

- 1. Center for Drug Evaluation and Research, Food and Drug Administration, U.S. Department of Health and Human Services. (2013, June). *Guidance for industry: Human immunodeficiency virus-1 infection: Developing antiretroviral drugs for treatment*. Retrieved from <a href="http://www.fda.gov/drugs/guidancecomplianceregulatoryinformation/guidances/ucm355239.htm">http://www.fda.gov/drugs/guidancecomplianceregulatoryinformation/guidances/ucm355239.htm</a>.
- 2. International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use. (1995, November 30). *ICH E3: Structure and content of clinical study reports*. Retrieved from http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html.

6. Proposed Summary Listings and Tables

# ATTACHMENT TaiMed Biologics, Inc.

## **Protocol TMB-311**

A Phase 3, Multicenter, Expanded Access Study of Ibalizumab Plus an Optimized Background Regimen (OBR) in Treatment-Experienced Patients Infected With Multi-Drug Resistant (MDR) HIV-1

# **Mock Statistical Listings**

November 9, 2017 Final Version 2

TaiMed Biologics, Inc 2 Executive Circle, Suite 280 Irvine, CA 92614

Prepared By:
Ken Gerald, PhD
Director of Biostatistics
and
Jennifer Fulton, MS
Biostatistician

Westat 5615 Kirby Drive, Suite 710 Houston, TX 77005

**CONFIDENTIAL** 

# **Notes Applicable to All Listings**

#### General Programming Notes:

- 1. There are a few listings that might fit as they are or might have to be split once we see the output with actual data.
- 2. All listings should start with and be sorted by Patient ID (concatenation of site number and patient number) and then visit date as appropriate.
- 3. If columns with specific text should be widened due to the amount of text, it is up to the programmer's discretion. However, please keep to the industry standard margin of 1 inch on bottom and sides and 1.25 inches on the top. Font is Courier New 8 point.
- 4. For all dates used, character format dates to capture partial dates. Use dashes where a month or day is missing. If entire date is missing just leave blank. i.e., JAN2011 or 01-2011.
- 5. If a programming note appears on the mock listing indicating that the footnote should appear only on the first page, this means the first page of output contains all footnotes and ONLY footnotes. All subsequent pages contain data with one footnote that says "Refer to page 1 for footnotes".
- 6. Some of the mock tables display numbers rather than x's. The numbers are meaningless and are for example only. Where visit names are displayed in tables, these are examples as well. Correct visit names for the TMB-311 study should be displayed in the actual output.
- 7. Each listing should include all applicable data, even if only a subset of the full set of treatment groups is displayed in the mocks. And unlike the tables and graphs, the listings should also include the 2 PI-IND rollover patients.
- 8. Sort each listing by Treatment and then Patient ID where applicable.

Listing 16.2.1.1

Patient Disposition

| Treatment | Patient<br>ID Sc | reened | ITT<br>Population<br>[1] | SAF<br>Population<br>[2] |
|---|---|---|---|---|
| C1:301/800mg | 311-XX-XXX | YES | YES | YES |
| C1:202/800mg | 311-XX-XXX | YES | YES | YES |
| C1:202/2000mg | 311-XX-XXX | YES | YES | YES |
| C2:800mg | 311-XX-XXX | YES | YE: | S YES |

<sup>[1]</sup>Intent-to-Treat (ITT) Population consists of all patients enrolled into the study.

Programming note: Add the mITT population if analyst decides it is needed later.

Westat (Created on DDMMYYYY)
S:\TMB311\DA\SAS\L PATDISP.SAS

<sup>[2]</sup>Safety (SAF) Population consists of patients receiving at least one partial dose of study drug.

Listing 16.2.1.2 Study Discontinuation

| Treatment | Patient<br>ID | Study<br>Discontinuation<br>Date | Date of<br>Last<br>Treatment | Completed<br>Study<br>Treatment | Reason for<br>Treatment<br>Discontinuation | Completed<br>Study | Reason for Study<br>Discontinuation | Death<br>Date |
|---|---|---|---|---|---|---|---|---|
| C2:800mg | 311-XX-XX | x 20161101 | 20161004 | NO | CONSENT WITHDRAWN OR<br>VOLUNTARY WITHDRAWAL | NO | CONSENT WITHDRAWN OR<br>VOLUNTARY WITHDRAWAL | |
| C2:800mg | :800mg 311-XX-XXX 20160920 | | | | ADVERSE EVENT-SEVERE DRUG<br>RASH AND FEVER OF 1<br>WEEK. | NO | ADVERSE EVENT-SEVERE DRUG<br>RASH AND FEVER OF 1<br>WEEK. | |
| C1:202/2000mg | 311-XX-XX | x 20160517 | 20160421 | NO | INVESTIGATORS DECISION-INVESTIGATORS DECISION | NO | INVESTIGATORS DECISION-LACK OF CLINICAL PROGRESSION | |
| C2:800mg | :800mg 311-XX-XXX 2016110 | | 20160810 | NO | INVESTIGATORS DECISION-SUBJECT NEVER CAME TO FOLOOW UP VISIT BECAUSE NEVER RECOVERED FROM PCP | NO | INVESTIGATORS DECISION-SUBJECT NEVER CAME TO F/UP VISIT BECAUSE NEVER RECOVERED FROM PNEUMONIA | |
| C1:301/800mg | 1/800mg 311-XX-XXX 20160728 20160728 NO | | CONSENT WITHDRAWN OR NO VOLUNTARY WITHDRAWAL | | CONSENT WITHDRAWN OR VOLUNTARY WITHDRAWAL | | | |
| C1:202/800mg | 311-XX-XX | X 20161004 | 20160720 | NO | ADVERSE EVENT-SUBJECT<br>DECEASED AS RESULT OF<br>TRAUMA DURING ACCIDENTAL<br>FALL | NO | ADVERSE EVENT-SUBJECT<br>DECEASED AS RESULT OF<br>TRAUMA DURING ACCIDENTAL<br>FALL | 20161 |

Westat (Created on DDMMMYYYY)
S:\TMB311\DA\SAS\L\_DISCRSN.SAS

Listing 16.2.2.1
Text of Inclusion and Exclusion

| Criterion<br>Type | Criterion<br>Number | Criterion Text |
|---|---|---|
| Inclusion | 1 | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | 2 | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| | 9 | |
| Exclusion | 1 | $ \begin{array}{c} x \\ x \\ \end{array} $ |
| | 2 | |
| | 12 | |

TaiMed Biologics, Inc. TMB-311

#### Listing 16.2.2.2 Protocol Violations

| Treatment | Patient | | Protocol | Details | Approval | Date of |
|---|---|---|---|---|---|---|
| | ID | Visit | Violation Code | of Violation | Obtained | Approval |
| C1:202/800mg | 311-XX-XXX | XXXXXX | XXX | XXXXXXXXXX | Yes/No | DDMONYYYY |
| C1:202/2000mg | 311-XX-XXX | XXXXXX | XXX | XXXXXXXXX | Yes/No | DDMONYYYY |

Westat (Created on DDMMMYYYY)
S:\TMB311\DA\SAS\L\_PROTVIOS.SAS

TaiMed Biologics, Inc. TMB-311

## Listing 16.2.2.3 Protocol Deviations

| Treatment | Patient | | Protocol | Details of | Approval | Date of |
|---|---|---|---|---|---|---|
| | ID | Visit | Deviation Code | Deviation | Obtained | Approval |
| C1:202/2000mg | 311-XX-XXX | XXXXXX | XXX | XXXXXXXXXX | Yes/No | DDMONYYYY |
| C2:800mg | 311-XX-XXX | XXXXXX | XXX | XXXXXXXXX | Yes/No | DDMONYYYY |

Westat (Created on DDMMMYYYY)
S:\TMB311\DA\SAS\L\_PROTDEV.SAS

Listing 16.2.2.4 Inclusion/Exclusion Criteria Violations/Deviations

| | | | Time of | | | | |
|---|---|---|---|---|---|---|---|
| | | Date of | Informed | Subject be | Criterion | | |
| | Patient | Informed | Consent | Enrolled in | Type and | Approval | Date of |
| Treatment | ID | Consent | (hh:mm) | Study | Number [1] | Obtained | Approval |
| C1:301/800mg | 311-XX-XXX | DDMONYYYY | XX:XX | Yes/No | EXC XXX/INC | Yes/No | DDMONYYYY |
| | 211-VV-VVV | DDMONIIII | AA • AA | | XXX | | |
| C1:202/800mg | 311-XX-XXX | DDMONYYYY | XX:XX | Yes/No | EXC XXX/INC | Yes/No | DDMONYYYY |
| | DII VV-VVV | DDMONIII | ΛΛ • ΛΛ | | XXX | | |

[1] Refer to Listing 16.2.2.1 for text.

Westat (Created on DDMMMYYYY)
S:\TMB311\DA\SAS\L\_INCEXLVIOS.SAS

Listing 16.2.4.1.1

Demographic Characteristics

| Treatment | Patient ID | Date of Birth | Age (years) [1] | Ethnicity | Race | Sex |
|---|---|---|---|---|---|---|
| C1:301/800mg | 311-XX-XXX | 1962-01-22 | 54 | NOT HISPANIC OR LATINO | BLACK OR AFRICAN AMERICAN | М |
| C1:202/800mg | 311-XX-XXX | 1954-11-26 | 61 | NOT HISPANIC OR LATINO | WHITE | М |
| C2:800mg | 311-XX-XXX | 1988-02-11 | 28 | NOT HISPANIC OR LATINO | BLACK OR AFRICAN AMERICAN | М |
| C1:2000mg | 311-XX-XXX | 1960-12-16 | 55 | HISPANIC OR LATINO | UNKNOWN | М |
| C1:301/800mg | 311-XX-XXX | 1962-11-15 | 53 | NOT HISPANIC OR LATINO | WHITE | М |
| C2:800mg | 311-XX-XXX | 1966-04-21 | 50 | NOT HISPANIC OR LATINO | WHITE | М |

 $\label{lem:westat} \begin{tabular}{ll} We stat & (Created on DDMMMYYYY) \\ S:$TMB311$DA$SAS$L_DEMOG.SAS \\ \end{tabular}$ 

<sup>[1]</sup> Age = Age at Screening.

Listing 16.2.4.1.2
Demographic Characteristics
Screen Failures

| Treatment | Patient ID | Date of Birth | Age (years) [1] | Ethnicity | Race | Sex |
|---|---|---|---|---|---|---|
| SCREEN FAILURE | 311-XX-XXX | 1962-01-22 | 54 | NOT HISPANIC OR LATINO | BLACK OR AFRICAN AMERICAN | М |
| SCREEN FAILURE | 311-XX-XXX | 1954-11-26 | 61 | NOT HISPANIC OR LATINO | WHITE | М |
| SCREEN FAILURE | 311-XX-XXX | 1988-02-11 | 28 | NOT HISPANIC OR LATINO | BLACK OR AFRICAN AMERICAN | М |
| SCREEN FAILURE | 311-XX-XXX | 1960-12-16 | 55 | HISPANIC OR LATINO | UNKNOWN | М |
| SCREEN FAILURE | 311-XX-XXX | 1962-11-15 | 53 | NOT HISPANIC OR LATINO | WHITE | М |
| SCREEN FAILURE | 311-XX-XXX | 1966-04-21 | 50 | NOT HISPANIC OR LATINO | WHITE | М |

Westat (Created on DDMMMYYYY)
S:\TMB311\DA\SAS\L\_DEMOGSCR.SAS

<sup>[1]</sup> Age = Age at Screening.

## Listing 16.2.4.2 Medical History

| Treatment | Patient<br>ID | Medical Condition/Surgery | Start Date | Stop Date |
|---|---|---|---|---|
| C1:301/800mg | 311-XX-XXX | xxxxxxxxxxxx | DDMONYYYY | DDMONYYYY or ONGOING |
| C2:800mg | 311-xx-xxx | xxxxxxxxxxxx | DDMONYYYY | DDMONYYYY or ONGOING |

#### Listing 16.2.5.1 Study Drug Administration

| | Patient | | Visit | | Start Time S | | : | Infusion | Starting<br>Volume | Ending | Was entire | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Patient | | VISIT | | or infusion | infusion | | infusion | volume | Volume | dose | Reason if No or |
| Treatment | ID | Visit | Date | Dose (mg) | (hh:mm) | (hh:mm) | Infusion Site | Side | (ml) | (ml) | delivered? | Interrupted |
| C1:301/800m | 311-XX-XXX | xxxxxxx | DDMONYYYY | 2000/800 | xx:xx | XX:XX | Cephalic Vein/Other<br>Vein | Left/ | xxx | xxx | Yes/No/Yes w/<br>Interruption | xxxxxxxx |
| | | xxxxxx | DDMONYYYY | 2000/800 | XX:XX | XX:XX | Cephalic Vein/Other | Right | | | Yes/No/Yes w/ | |
| | | | | | | | Vein | Left/ | xxx | xxx | Interruption | |
| | | | | | | | | Right | | | | |
| C2:800mg | 311-xx-xxx | xxxxxxx | DDMONYYYY | 2000/800 | XX:XX | xx:xx | Cephalic Vein/Other<br>Vein | Left/ | xxx | xxx | Yes/No/Yes w/<br>Interruption | xxxxxxxx |
| | | | | | | | | Right | | | | |

Listing 16.2.5.2 ART Exposure

| Treatment | Patient<br>ID | Medication | Standardized<br>Medication<br>Name [1] | Indication | Start Date | Stop Date | Dose | Unit | Route | Frequency |
|---|---|---|---|---|---|---|---|---|---|---|
| C1:202/2000<br>mg | 311-XX-<br>XXX | xxxxxxx | xxxxxxx | xxxxxxx | DDMONYYYY | DDMONYYYY<br>Or ONGOING | xxxx | xxxx | xxxxx | xx |
| C2:800mg | 311-xx-<br>xxx | xxxxxxx | xxxxxxx | xxxxxxx | DDMONYYYY | DDMONYYYY<br>Or ONGOING | xxxx | xxxx | xxxxx | хх |

<sup>[1]</sup> Medications were coded with WHO Drug Dictionary Version March, 2014.

Westat (Created on DDMMMYYYY)
S:\TMB311\DA\SAS\L\_ARTEXP.SAS

Listing 16.2.5.3 Previous and Concomitant Medications

| Treatment | Patient ID | Medication | Standardized<br>Medication<br>Name [1] | Indication | Start Date | Stop Date | Dose | Unit | Route | Frequency |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | DDMONYYYY | DDMONYYYY | | | | |
| C1:202/800 mg | 311-xx-xxx | xxxxxxx | xxxxxxx | xxxxxxx | | Or ONGOING | xxxx | xxxx | xxxxx | xx |
| | | | | | | DDMONYYYY | | | | |
| C2:800mg | 311-XX-XXX | xxxxxxx | xxxxxxx | xxxxxxx | DDMONYYYY | Or ONGOING | xxxx | xxxx | xxxxx | xx |

<sup>[1]</sup> Medications were coded with WHO Drug Dictionary Version March, 2014.

Westat (Created on DDMMMYYYY)
S:\TMB311\DA\SAS\L\_CONMED.SAS

## Listing 16.2.5.4 Concomitant Procedures

| | Patient<br>ID | Procedure | Procedure Date | Reason |
|--------------|---------------|-----------|----------------|---------|
| Treatment | | | | |
| C1:301/800mg | 311-XX-XXX | xxxxxxx | DDMONYYYY | xxxxxxx |
| C2:800mg | 311-xx-xxx | XXXXXXX | DDMONYYYY | xxxxxxx |

Westat (Created on DDMMMYYYY)
S:\TMB311\DA\SAS\L\_CONPROCS.SAS

Listing 16.2.5.5 Optimized Background Regimen (OBR)

| Treatment | Patient<br>ID | Medication | Standardized<br>Medication<br>Name [1] | Indication | Start Date | Stop Date | Dose | Unit | Route | Frequency | Reason<br>for<br>Change |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | DDMONYYYY | DDMONYYYY | | | | | |
| C1:301/800m<br>g | 311-XX-<br>XXX | xxxxxxx | xxxxxxx | xxxxxxx | | Or ONGOING | xxxx | xxxx | xxxxx | xx | xxx |
| | 311-xx- | | | | | DDMONYYYY | | | | | |
| C2:800mg | XXX | xxxxxxx | xxxxxxx | xxxxxxx | DDMONYYYY | Or ONGOING | xxxx | xxxx | xxxxx | xx | xxx |

<sup>[1]</sup> Medications were coded with WHO Drug Dictionary Version March, 2014.

Westat (Created on DDMMMYYYY)
S:\TMB311\DA\SAS\L\_OBR.SAS

Listing 16.2.5.6 Optimized Background Regimen (OBR) Adherence

| | Patient | | | Has the patient taken all required doses of OBR | |
|---|---|---|---|---|---|
| Treatment | ID | Visit | Visit Date | since the last visit? | If No Explain |
| C1:202/800mg | :202/800mg 311-XX-XXX XXXXX DDMONYYYY | | DDMONYYYY | YES/NO | xxxxxxxxxx |
| C1:202/2000mg | | XXXX | DDMONYYYY | YES/NO | xxxxxxxxxxx |

Westat (Created on DDMMMYYYY) S:\TMB311\DA\SAS\L\_OBRADHER.SAS

Listing 16.2.6.1 Post-Injection Observation

| | | | | | Start Time of<br>Observation | End Time of<br>Observation | |
|---|---|---|---|---|---|---|---|
| Treatment | Patient<br>ID | Visit | Visit Date | Observed After<br>Study Drug | (hh:mm) | (hh:mm) | Comments |
| C1:301/800mg | 311-xx-xxx | xxx | DDMONYYYY | YES/NO | xx:xx | XX:XX | xxxxxxxxxxxxxx |
| C2:800mg | 311-xx-xxx | xxx | DDMONYYYY | YES/NO | xx:xx | xx:xx | xxxxxxxxxxxxxxx |

Westat (Created on DDMMMYYYY)
S:\TMB311\DA\SAS\L\_POSTINJECT.SAS

#### Listing 16.2.6.2 CD4+ Cell Count (cells/mm^3)

# Unimputed Original Values Imputed with LOCF [5]

| Treatment | Patient<br>ID | Visit<br>[1] | Visit Date<br>(Study Day) | CD4+ Cell<br>Count<br>(cells/mm^3)<br>[2] | CD4+ Cell Count<br>Change from<br>Baseline (%) | Toxicity [4] | CD4+ Cell<br>Count (cells/mm^3)<br>[2] | CD4+ Cell Count<br>Change from<br>Baseline (%) |
|---|---|---|---|---|---|---|---|---|
| C1:301/800mg | 311-XX-XXX | XXXXXXX | DDMONYYYY (XX) | XXX* | XXXX | XXXX | XXX* | XXXX |
| C2:800mg | 311-XX-XXX | XXXXXXX | DDMONYYYY (XX) | XXX | XXXX | XXXX | XXX | XXXX |

[1] EOS=End of Study visit conducted at Week 174 (for TMB-301 rollovers)/Week 150 (for all other patients).

[2]\*=below 200 cells/mm^3

[3]Calculated as (visit value - baseline)/baseline\*100%

[4]Toxicity is defined as 2 consecutive laboratory results, at least 14 days apart, with a CD4+ cell count below 200 cells/mm3 that also represents a 50% reduction from the baseline CD4+ cell count.

[5] Missing values are imputed using the Last Observation Carried Forward (LOCF) method.e

Westat (Created on DDMMMYYYY)
S:\TMB311\DA\SAS\L\_CD4.SAS
# Listing 16.2.6.5 Viral Load

Chg from Chg from Chg from Treatment Date Viral Load Baseline HIV-1 RNA Viral Load Baseline HIV-1 RNA

Patient Visit Visit Date (Study Day) (log10 (log10 (cp/mL) (log10 (cp/mL) Treatment ID [2] (Study Day) [3] cp/mL) cp/mL) [5] cp/mL) [5]

| DAY 0 | 2016-08-22 20 | 16-08-10 (159) 1 | .0 TND** | 1.0 | TND** |
|---|---|---|---|---|---|
| C1:301/800mg 311-XX | -XXX DAY 14 | | 4.9 | 0.0 73 | 700 |
| WEEK 12 | ! | | 4.9 0.0 737 | 00 | |
| WEEK 16 | j | | 4.9 0.0 737 | 00 | |
| WEEK 12 | 2016-11-14 (84) | 2016-10-31 (245) | 1.3 -3.6 TD** | 1.3 | -3.6 TD** |
| WEEK 20 | ) | | 4.9 0.0 737 | 00 | |
| WEEK 24 | ļ | | 4.9 0.0 737 | 00 | |
| WEEK 24 | 2017-02-06 (168) | 2017-01-23 (329) | 1.0 -3.9 TND** | 1.0 | -3.9 TND** |
| 311-XX-XXX DA | AY 0 2016-09-07 | 2016-08-24 (154) | ) 1.3 TD** | 1.3 | TD** |
| DAY 14 | | | 3.8 0.0 6530 | | |
| WEEK 12 | <u>!</u> | | 3.8 0.0 653 | ) | |
| WEEK 16 | 5 | | 3.8 0.0 653 | 0 | |
| WEEK 12 | 2016-12-01 (352) | 2016-11-17 (513) | 1.0 -2.8 TND** | 1.0 | -2.8 TND** |
| WEEK 20 | ) | | 3.8 0.0 653 | ) | |
| WEEK 24 | ļ | | 3.8 0.0 653 | 0 | |
| WEEK 24 | 2017-02-23 (436) | 2017-02-10 (598) | 1.0 -2.8 TND** | 1.0 | -2.8 TND** |

<sup>[1]</sup> EOS=End of Study visit conducted at Week 174 (for TMB-301 rollovers)/Week 150 (for all other patients).

(Continued)

<sup>[2]</sup> Visits are assigned based on study day using the windows defined in the statistical analysis plan.

<sup>[3]</sup> Last treatment prior to viral load measurement.

<sup>[4]</sup> Viral Load results are imputed based on MEF (Missing Equals Failure). This means null viral load results are replaced with the baseline value such that Change from Baseline=0 and the result is a failure. Also all records following a CONFIRMED virologic failure are set to failure.

<sup>[5] \*=</sup>below 400 copies/mL; \*\*=below 50 copies/mL. HIV-1 RNA level results below level of quantitation are coded as target detected (TD) or target not detected (TND).

#### At EOS

| Treatment | Patient<br>ID | Visit<br>[1] | Visit Date<br>(Study Day) | | | |
|---|---|---|---|---|---|---|
| | | | | Virologic Outcome [2] | Virologic Failure [3] | Virologic Success [4] |
| C1:301/800mg | 311-XX-XXX | XXXXXXX | DDMONYYYY<br>(XX) | XX | XXXXXXX | XXXXXXX |
| C2:800mg | 311-XX-XXX | XXXXXXX | DDMONYYYY<br>(XX) | XX | XXXXXXX | XXXXXXX |

[1] Visits are assigned based on study day using the windows defined in the statistical analysis plan.

[2] Per the Snapshot Approach:

1=Virologic success (=0.5 log copies/mL drop from Baseline in viral load)

2a=(<0.5 log copies/mL drop from Baseline in viral load)

2b=Discontinued because of virologic failure

2c=Discontinued because of other reasons and drop from baseline in viral load at the time of discontinuation was <0.5 log copies/mL

### 2d=OBR changed

## 3a=Discontinued because of AE or death

3b=Discontinued because of other reasons and drop from baseline in viral load at the time of discontinuation was >=0.5 log copies/mL

# 3c=Missing data during the window but on study

[3] Failure to achieve/maintain response=Patient does not have >=0.5 log10 decline from baseline(BL) by Week 12 on study drug OR patient has a 0.5 log10 decline from BL prior to Week 12 but fails to maintain the 0.5 log10 decline from BL with a <1 log10 increase from nadir on any two consecutive scheduled efficacy assessments after Week 12.

Rebound=Patient has a >=0.5 log10 decline from BL by Week 12 that is maintained but viral load remains >=50 copies (not suppressed), followed by >=1 log10 increase from nadir at two consecutive scheduled visits any time after the primary endpoint.

Breakthrough=Patient has suppressed viral load (< 50 copies) at any time after primary endpoint followed by >=200 copies at two consecutive scheduled efficacy assessments.

[4]Suboptimal Response=Patient has a 0.5 log10 decline but does not suppress (<50 copies) at any time after primary endpoint; Virologic Suppression=Patient has a 0.5 log10 decline and does suppress (<50 copies) at any time after primary endpoint

Programming note: See footnotes (values to the left of the =) to indicate what values will be displayed in the listing.

Westat (Created on DDMMMYYYY)
S:\TMB311\DA\SAS\L VLOUTCOMES.SAS

# Listing 16.2.6.7 Patients with Virologic Failure

### Patient ID

| Treatment | | Visit | Visit<br>Date | Viral Load<br>(log <sub>10</sub> copies/mL) | Change from<br>Baseline |
|---|---|---|---|---|---|
| C1:301/800mg | 311-XX-XXX | XXX | DDMONYYYY | XXX | XXX |
| C1:800 MG | 311-XX-XXX | XXX | DDMONYYYY | XXX | XXX |

Note: Virologic failure is defined as two consecutive measurements of less than a 0.5 log10 decline from the Baseline viral load. For the Cohort 2 and TMB-301 rollover patients, virologic failure will not be assessed prior to 24 weeks on study drug. For the TMB-202 rollover patients, virologic failure will not be assessed prior to the start of the TMB-311 study period.

Westat (Created on DDMMMYYYY)
S:\TMB311\DA\SAS\L VLFAIL.SAS

Listing 16.2.7.1
Adverse Events

| | | System | | Adverse | | | | | Sev. | | | Action | | Class |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Patient<br>ID | Organ<br>Class | Preferred<br>Term[1] | Event<br>Verbatim | TEAE<br>[2] | | art Date<br>idy Day) | Stop Date<br>(Study Day) | /Grade<br>[3] | SAE | Caus.<br>[4] | Taken<br>[5] | Outcm. [6] | C<br>AE |
| | | | | · | | | | | | | | | | |
| C1:301/800mg | 311-XX-XXX | MUSCULOSKELETAL AND CONNECTIVE TISSUE | ARTHRALGIA | MILD PAIN (I<br>TO FALL AT | OUE | Y | 20160923<br>(283) | 20161010 | ) 1 | | N 0 | | 0 1 | 1 |
| C2:800mg | 311-XX-XXX | NERVOUS SYSTEM<br>DISORDERS | HEADACHE | WORSENING<br>HEADACHES | | Y | 20160516 | 20160524<br>(11) | 2 | | N 0 | | 0 | 1 |
| | | INVESTIGATIONS | BREATH SOUNDS<br>ABNORMAL | DECREASED<br>BREATH SOUNI | os | Y | 20160520<br>(7) | 20160609<br>(27) | ) 1 | | N 0 | | 0 | 1 |
| C1:202/2000mg | 311-XX-XXX | RENAL AND URINARY<br>DISORDERS | POLLAKIURIA | URINARY<br>FREQUENCY | | Y | 20161005<br>(208) | | 2 | | N 0 | | 1 : | 3 |
| C1:202/800mg | 311-XX-XXX | SKIN AND<br>SUBCUTANEOUS TISSUE<br>DISORDERS | RASH<br>MACULO-PAPU-<br>LAR | MACULOPAPULA<br>RASH ON<br>EXTREMITIES | AR | Y | 20170119<br>(349) | 20170214<br>(375) | 1 2 | | N 1 | | 1 : | 1 |

Westat (Created on DDMMMYYYY)
S:\TMB311\DA\SAS\L AE.SAS

<sup>[1]</sup> Adverse events are coded using MedDRA Version 17.0.

<sup>[2]</sup> A treatment-emergent AE (TEAE) is defined as any event not present before exposure to study drug or any event already present that worsens in either intensity or frequency following exposure to study drug. AEs with missing start dates, but with stop dates either overlapping into the dosing period or missing, will be considered TEAEs

<sup>[3]</sup> Severity/Grade: 1=Mild, 2=Moderate, 3=Severe, 4=Potentially Life Threatening, 5=Death

<sup>[4]</sup> Causality: 0=Unrelated, 1=Possible, 2=Probable, 3=Definite

<sup>[5]</sup> Action Taken: 0=None, 1=Medication Given, 2=Non-Medication Therapy, 3=Suspended Study Drug, 4=Permanently Discontinued Study Drug, 99=Other

<sup>[6]</sup> Outcome: 1=Resolved, 2=Resolved w/sequelae, 3=Ongoing, 4=Worsened, 5=Death, 7=Chronic/Stable, 98=Unknown

Listing 16.2.7.2 Serious Adverse Events

| | | System | | Adverse | | | | Sev. | | | Action | | Class |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Patient<br>ID | Organ<br>Class | Preferred<br>Term[1] | Event<br>Verbatim | TEAE<br>[2] | Start Date<br>(Study Day) | Stop Date<br>(Study Day) | /Grade<br>[3] | SAE | Caus.<br>[4] | Taken<br>[5] | Outcm.<br>[6] | C<br>AE |
| C2:800mg | 311-XX-XXX | INVESTIGATIONS | BLOOD<br>POTASSIUM<br>DECREASED | LOW SERUM<br>POTASSIUM | Y | 20161116 (187) | 20161118 (189) | 3 | Y | 0 | 1,99 | 1 | |
| C1:301/800mg | 311-XX-XXX | INFECTIONS AND INFESTATIONS | CELLULITIS | FACE<br>CELLULITIS | Y | 20161017<br>(153) | 20161101 (168) | 2 | Y | 0 | 1,99 | 7 | |
| C1:202/2000m | g 311-XX-XXX | NEOPLASMS BENIGN,<br>MALIGNANT AND<br>UNSPECIFIED (INCL<br>CYSTS AND POLYPS) | TONSIL CANCER<br>METASTATIC | METASTATIC SQUAMOUS CEL CARCINOMA OF THE RIGHT TONSIL | Y<br>L | 20161130 (190) | | 4 | Y | 0 | 0 | 3 | |
| C1:202/800mg | 311-XX-XXX | NEOPLASMS BENIGN,<br>MALIGNANT AND<br>UNSPECIFIED (INCL<br>CYSTS AND POLYPS) | TONSIL CANCER<br>METASTATIC | METASTATIC SQUAMOUS CEL CARCINOMA OF THE RIGHT TONSIL | Y<br>L | 20170203<br>(255) | 20170204<br>(256) | 4 | Y | 0 | 1 | 4 | |
| | | NEOPLASMS BENIGN,<br>MALIGNANT AND<br>UNSPECIFIED (INCL<br>CYSTS AND POLYPS) | TONSIL CANCER<br>METASTATIC | METASTATIC<br>SQUAMOUS CEL<br>CARCINOMA OF<br>THE RIGHT | Y<br>L | 20170205<br>(257) | 20170205<br>(257) | 5 | Y | 0 | 1 | 5 | |

<sup>[1]</sup> Adverse events are coded using MedDRA Version 17.0.

Westat (Created on DDMMMYYYY)

<sup>[2]</sup> A treatment-emergent AE (TEAE) is defined as any event not present before exposure to study drug or any event already present that worsens in either intensity or frequency following exposure to study drug. AEs with missing start dates, but with stop dates either overlapping into the dosing period or missing, will be considered TEAEs.

<sup>[3]</sup> Severity/Grade: 1=Mild, 2=Moderate, 3=Severe, 4=Potentially Life Threatening, 5=Death

<sup>[4]</sup> Causality: 0=Unrelated, 1=Possible, 2=Probable, 3=Definite

<sup>[5]</sup> Action Taken: 0=None, 1=Medication Given, 2=Non-Medication Therapy, 3=Suspended Study Drug, 4=Permanently Discontinued Study Drug, 99=Other

<sup>[6]</sup> Outcome: 1=Resolved, 2=Resolved w/sequelae, 3=Ongoing, 4=Worsened, 5=Death, 7=Chronic/Stable, 98=Unknown

Listing 16.2.7.3

Adverse Events Leading to Study Discontinuation or Death

| | | System | | Adverse | | | | Sev. | | | Action | | Class |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | Patient<br>ID | Organ<br>Class | Preferred Term[1] | Event<br>Verbatim | TEAE<br>[2] | Start Date<br>(Study Day) | Stop Date<br>(Study Day) | /Grade<br>[3] | SAE | Caus.<br>[4] | Taken<br>[5] | Outcm. [6] | C<br>AE |
| | | | | | [2] | | (Seday Bay) | [9] | | | [9] | | |
| C1:2000mg | 311-XX-XXX I | NEOPLASMS BENIGN,<br>MALIGNANT AND<br>UNSPECIFIED (INCL<br>CYSTS AND POLYPS) | TONSIL CANCER<br>METASTATIC | METASTATIC<br>SQUAMOUS CELL<br>CARCINOMA OF<br>THE RIGHT<br>TONSIL | Y | 20170205<br>(257) | 20170205<br>(257) | 5 | Y | 0 | 1 | 5 | |
| C1:301/800mg | g 311-XX-XXX | GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS | PYREXIA | FEVER | Y | 20160830<br>(7) | 20160901 (9) | 3 | N | 1 | 1,4 | 1 | |
| C2:800mg | 311-XX-XXX | INFECTIONS AND INFESTATIONS | SEPSIS | SEPSIS<br>SECONDARY TO<br>NEUTROPENIA | Y | 20160901<br>(93) | 20161114<br>(167) | 5 | Y | 0 | 1,4 | 5 | YES |
| C1:202/800mç | g 311-XX-XXX | INJURY, POISONING<br>AND PROCEDURAL<br>COMPLICATIONS | INJURY | TRAUMA FROM<br>FALL | Y | 20161001<br>(157) | 20161001<br>(157) | 5 | Y | 0 | 4 | 5 | |

<sup>[1]</sup> Adverse events are coded using MedDRA Version 17.0.

Westat (Created on DDMMMYYY)
S:\TMB311\DA\SAS\L AEDISCDTH.SAS

<sup>[2]</sup> A treatment-emergent AE (TEAE) is defined as any event not present before exposure to study drug or any event already present that worsens in either intensity or frequency following exposure to study drug. AEs with missing start dates, but with stop dates either overlapping into the dosing period or missing, will be considered TEAEs

<sup>[3]</sup> Severity/Grade: 1=Mild, 2=Moderate, 3=Severe, 4=Potentially Life Threatening, 5=Death

<sup>[4]</sup> Causality: 0=Unrelated, 1=Possible, 2=Probable, 3=Definite

<sup>[5]</sup> Action Taken: 0=None, 1=Medication Given, 2=Non-Medication Therapy, 3=Suspended Study Drug, 4=Permanently Discontinued Study Drug, 99=Other

<sup>[6]</sup> Outcome: 1=Resolved, 2=Resolved w/sequelae, 3=Ongoing, 4=Worsened, 5=Death, 7=Chronic/Stable, 98=Unknown

Listing 16.2.8.1.1 Clinical Laboratory Test Hematology

| Treatment | Patient<br>ID | Visit [1] | Date of Sample<br>(Study Day) | Test | Result<br>(L/H)[2] | Unit | Lower<br>Limit of<br>Normal | Upper<br>Limit of<br>Normal | Potentially<br>Clinically<br>Significant[3 |
|---|---|---|---|---|---|---|---|---|---|
| C1:301/800mg | 311-XX-XXX | XXXXXXXXX | 2016-03-04 (-172) | Basophils | 0 | 10^9/L | 0 | 0.2 | |
| , | | | , | Basophils/Total Cells | 0 | % | 0 | 2 | |
| | | | | Eosinophils | 0.02 | 10^9/L | 0 | 0.57 | |
| | | | | Eosinophils/Total Cells | 1 | - · · · / - · | 0 | 6.8 | |
| | | | | Hematocrit | 0.31(L) | Proport- | 0.39 | 0.54 | YES |
| C1:800mg | 311-XX-XXX | XXXXXXXXX | 2016-11-14 (84) | Hemoglobin | 106(L) | a/T | 127 | 181 | YES |
| | | | , | Leukocytes | 1.62(L) | 10^9/L | 3.8 | 10.7 | YES |
| | | | | Lymphocytes | 0.6(L) | 10^9/L | 0.91 | 4.28 | YES |
| | | | | Lymphocytes/Total Cells | 37 | 8 | 15.4 | 48.5 | |
| | | | | Monocytes | 0.16 | 10^9/L | 0.12 | 0.92 | |
| | | | | Monocytes/Total Cells | 10 | 8 | 2.6 | 10.1 | |
| | | | | Neutrophils | 0.84(L) | 10^9/L | 1.96 | 7.23 | YES |
| | | | | Neutrophils/Total Cells | 52 | 용 | 40.5 | 75 | |
| | | | | Platelets | 278 | 10^9/L | 140 | 400 | |
| C1:2000mg | 311-XX-XXX | XXXXXXXXX | 2016-11-14 (84) | Basophils | 0.08 | 10^9/L | 0 | 0.2 | |
| J. | | | | Basophils/Total Cells | 2.3(H) | 용 | 0 | 2 | YES |
| | | | | Eosinophils | 0.19 | 10^9/L | 0 | 0.57 | |
| | | | | Eosinophils/Total Cells | 5.5 | 용 | 0 | 6.8 | |
| | | | | Hematocrit | 0.39 | Proport- | 0.39 | 0.54 | |
| C2:800mg | 311-XX-XXX | XXXXXXXXX | 2016-11-14 (84) | Hemoglobin | 128 | g/L | 127 | 181 | |
| | | | | Leukocytes | 3.47(L) | 10^9/L | 3.8 | 10.7 | YES |
| | | | | Lymphocytes | 1.49 | 10^9/L | 0.91 | 4.28 | |
| | | | | Lymphocytes/Total Cells | 43 | 용 | 15.4 | 48.5 | |
| | | | | Monocytes | 0.34 | 10^9/L | 0.12 | 0.92 | |
| | | | | Monocytes/Total Cells | 9.7 | 8 | 2.6 | 10.1 | |
| | | | | Neutrophils | 1.37(L) | 10^9/L | 1.96 | 7.23 | YES |
| | | | | Neutrophils/Total Cells | 39.5(L) | 8 | 40.5 | 75 | YES |
| | | | | Platelets | 250 | 10^9/L | 140 | 400 | |

<sup>[1]</sup> For TMB301 Rollovers, BASELINE is the value recorded on Day 7 of the TMB-301 study. For TMB202 Rollovers, BASELINE is the value recorded on Day 0 of the TMB-202 study. Lab samples were not collected at the TMB-311 Screening for the Cohort 1 patients. EOS=End of Study visit conducted at Week 96.

<sup>[2]</sup> L = Below lower limit of normal; H = Above upper limit of normal.

<sup>[3]</sup> Potentially Clinically Significant is defined as having a result either below the lower limit of normal or above the upper limit of normal.

Listing 16.2.8.1.2
Clinical Laboratory Test
Chemistry

| Treatment | Patient<br>ID | Visit [1] | Date of Sample<br>(Study Day) | Test | Result<br>(L/H)[2] | Unit | Lower<br>Limit of<br>Normal | Upper<br>Limit of<br>Normal | Potentially<br>Clinically<br>Significant[3 |
|---|---|---|---|---|---|---|---|---|---|
| 1:301/800mg | 311-XX-XXX | XXXXXXX | 2016-03-04 (-172) | Alanine Aminotransferase | 21 | U/L | 6 | 43 | |
| <u> </u> | | | | Albumin | 36 | g/L | 33 | 49 | |
| | | | | Alkaline Phosphatase | 100 | Ū/L | 35 | 131 | |
| | | | | Amylase | 167(H) | U/L | 28 | 120 | YES |
| 1:202/800mg | 311-XX-XXX | XXXXXXX | 2016-11-14 (84) | Alanine Aminotransferase | 18 | U/L | 6 | 43 | |
| | | | | Albumin | 38 | g/L | 33 | 49 | |
| | | | | Alkaline Phosphatase | 131 | U/L | 35 | 131 | |
| | | | | Amylase | 158(H) | U/L | 28 | 120 | YES |
| | | | | Aspartate Aminotransferase | 20 | U/L | 11 | 36 | |
| 1:202/2000mg | 311-XX-XXX | XXXXXXXX | 2016-03-04 (-172) | Alanine Aminotransferase | 21 | U/L | 6 | 43 | |
| | | | | Albumin | 36 | g/L | 33 | 49 | |
| | | | | Alkaline Phosphatase | 100 | U/L | 35 | 131 | |
| | | | | Amylase | 167(H) | U/L | 28 | 120 | YES |
| 2:800mg | 311-XX-XXX | XXXXXXX | 2016-11-14 (84) | Alanine Aminotransferase | 18 | U/L | 6 | 43 | |
| | | | | Albumin | 38 | g/L | 33 | 49 | |
| | | | | Alkaline Phosphatase | 131 | U/L | 35 | 131 | |
| | | | | Amylase | 158(H) | U/L | 28 | 120 | YES |
| | | | | Aspartate Aminotransferase | 20 | U/L | 11 | 36 | |

<sup>[1]</sup> For TMB301 Rollovers, BASELINE is the value recorded on Day 7 of the TMB-301 study. For TMB202 Rollovers, BASELINE is the value recorded on Day 0 of the TMB-202 study. Lab samples were not collected at the TMB-311 Screening for the Cohort 1 patients. EOS=End of Study visit conducted at Week 96.

Westat (Created on DDMMMYYYY)
S:\TMB311\DA\SAS\L LABCHEM.SAS

<sup>[2]</sup> L = Below lower limit of normal; H = Above upper limit of normal.

<sup>[3]</sup> Potentially Clinically Significant is defined as having a result either below the lower limit of normal or above the upper limit of normal.

Listing 16.2.8.1.3 Clinical Laboratory Test Urinalysis

| Treatment | Patient<br>ID | Visit | Date of Sample<br>(Study Day) | Test | Unit | Result |
|---|---|---|---|---|---|---|
| C1:301/800mg | 311-XX-XXX | xxxxxxxx | 2016-03-04 (-172) | Calcium Oxalate Crystals<br>Hyaline Casts<br>Sediment Examination | /LPF | Present<br>2<br>Positive |
| | | XXXXXXX | 2016-11-14 (84) | Sediment Examination | | Positive |
| | | xxxxxxx | 2017-02-06 (168) | Sediment Examination | | Positive |
| C1:202/800mg | 311-XX-XXX | xxxxxxx | 2016-03-16 (92) | Mucous Threads | | Present |
| | | XXXXXXX | 2016-03-23 (99) | Calcium Oxalate Crystals<br>Sediment Examination | | Present<br>Positive |
| | | XXXXXXX | 2017-02-23 (436) | Amorphous Crystals<br>Sediment Examination | | Present<br>Positive |
| C2:800mg | 311-XX-XXX | xxxxxxx | 2016-04-07 (-37) | Sediment Examination | | Positive |
| | | XXXXXXXX | 2016-05-13 (0) | Sediment Examination | | Positive |
| | | XXXXXXX | 2016-05-20 (7) | Hyaline Casts<br>Sediment Examination | /LPF | 2<br>Positive |
| C1:202/2000mg | 311-XX-XXX | XXXXXXXX | 2016-03-11 (0) | Sediment Examination | | Negative |
| | | xxxxxxx | 2016-06-03 (84) | Calcium Oxalate Crystals<br>Mucous Threads<br>Sediment Examination | | Present<br>Present<br>Positive |
| | | XXXXXXX | 2016-08-25 (167) | Sediment Examination | | Negative |

EOS=End of Study visit conducted at Week 96.

Listing 16.2.8.1.4
Abnormal Laboratory Results

| Treatment | Patient<br>ID | Visit [1] | Date of Sample<br>(Study Day) | Category | Test | Result<br>(L/H)[2] | Unit | Lower<br>Limit of<br>Normal | Upper<br>Limit of<br>Normal | Potentially<br>Clinically<br>Significant[3] |
|---|---|---|---|---|---|---|---|---|---|---|
| C1:301/800mg | 311-XX-XXX | xxxxxxxx | 2016-03-04 (-172) | ) CHEMISTRY | Amylase | 167 (H) | U/L | 28 | 120 | YES |
| | | | | | Direct Bilirubin | 1(L) | umol/L | 2 | 7 | YES |
| | | | | HEMATOLOGY | Hematocrit | 0.31(L) | Proportion of 1 | 0.39 | 0.54 | YES |
| | | | | | Hemoglobin | 106(L) | g/L | 127 | 181 | YES |
| | | | | | Leukocytes | 1.62(L) | 10^9/L | 3.8 | 10.7 | YES |
| | | | | | Lymphocytes | 0.6(L) | 10^9/L | 0.91 | 4.28 | YES |
| | | | | | Neutrophils | 0.84(L) | 10^9/L | 1.96 | 7.23 | YES |
| C1:202/800mg | 311-XX-XXX | XXXXXXXXX | 2016-11-14 (84) | CHEMISTRY | Amylase | 158(H) | U/L | 28 | 120 | YES |
| | | | | | Bilirubin | 1.5(L) | umol/L | 3 | 21 | YES |
| | | | | | Direct Bilirubin | 1(L) | umol/L | 2 | 7 | YES |
| | | | | HEMATOLOGY | Basophils/Total<br>Cells | 2.3(H) | % | 0 | 2 | YES |
| | | | | | Leukocytes | 3.47(L) | 10^9/L | 3.8 | 10.7 | YES |
| | | | | | Neutrophils | 1.37(L) | 10^9/L | 1.96 | 7.23 | YES |
| | | | | | Neutrophils/Total<br>Cells | 39.5(L) | % | 40.5 | 75 | YES |
| C1:202/2000mg | 311-XX-XXX | XXXXXXXXX | 2017-02-06 (168) | CHEMISTRY | Amylase | 133(H) | U/L | 28 | 120 | YES |
| | | | | | Direct Bilirubin | 1(L) | umol/L | 2 | 7 | YES |
| | | | | HEMATOLOGY | Hematocrit | 0.37(L) | Proportion of 1 | 0.39 | 0.54 | YES |
| | | | | | Hemoglobin | 124(L) | g/L | 127 | 181 | YES |
| C2:800mg | 311-XX-XXX | XXXXXXXX | 2016-03-23 (99) | CHEMISTRY | Alanine<br>Aminotransferase | 68 (H) | U/L | 6 | 43 | YES |
| | | | | | Aspartate<br>Aminotransferase | 59(H) | U/L | 11 | 36 | YES |
| | | | | | Cholesterol | 3.03(L) | mmol/L | 4.53 | 7.71 | YES |
| | | | | | Creatine Kinase | 393 (H) | U/L | 39 | 308 | YES |

<sup>[1]</sup> For TMB301 Rollovers, BASELINE is the value recorded on Day 7 of the TMB-301 study. For TMB202 Rollovers, BASELINE is the value recorded on Day 0 of the TMB-202 study. Lab samples were not collected at the TMB-311 Screening for the Cohort 1 patients. EOS=End of Study visit conducted at Week 96.

Westat (Created on DDMMMYYYY)
S:\TMB311\DA\SAS\L LABABN.SAS

<sup>[2]</sup> L = Below lower limit of normal; H = Above upper limit of normal.

<sup>[3]</sup> Potentially Clinically Significant is defined as having a result either below the lower limit of normal or above the upper limit of normal.

Listing 16.2.8.1.5 Other Laboratory Results

| Treatment | Patient<br>ID | Visit [1] | Date of Sample<br>(Study Day) | Category | Test | Result<br>(L/H)[2] | Unit | Lower<br>Limit of<br>Normal | Upper<br>Limit of<br>Normal | Potentially<br>Clinically<br>Significant[3] |
|---|---|---|---|---|---|---|---|---|---|---|
| C1:301/800mg | 311-XX-XXX | x xxxxxxxx | 2016-03-04 ( | -172) CHEMISTRY | Amylase | 167(H) | U/L | 28 | 120 | YES |
| | | | | | Direct Bilirubin | 1(L) | umol/L | 2 | 7 | YES |
| | | | | HEMATOLOGY | Hematocrit | 0.31(L) | Proportion of 1 | 0.39 | 0.54 | YES |
| | | | | | Hemoglobin | 106(L) | g/L | 127 | 181 | YES |
| | | | | | Leukocytes | 1.62(L) | 10^9/L | 3.8 | 10.7 | YES |
| | | | | | Lymphocytes | 0.6(L) | 10^9/L | 0.91 | 4.28 | YES |
| | | | | | Neutrophils | 0.84(L) | 10^9/L | 1.96 | 7.23 | YES |
| C1:202/800mg | 311-XX-XXX | XXXXXXXXX | 2016-11-14 ( | 84) CHEMISTRY | Amylase | 158(H) | U/L | 28 | 120 | YES |
| | | | | | Bilirubin | 1.5(L) | umol/L | 3 | 21 | YES |
| | | | | | Direct Bilirubin | 1(L) | umol/L | 2 | 7 | YES |
| C1:202/2000mg | 311-XX-XXX | XXXXXXXXX | 2017-02-06 ( | 168) CHEMISTRY | Amylase | 133 (H) | U/L | 28 | 120 | YES |
| | | | | | Direct Bilirubin | 1(L) | umol/L | 2 | 7 | YES |
| | | | | HEMATOLOGY | Hematocrit | 0.37(L) | Proportion<br>of 1 | 0.39 | 0.54 | YES |

<sup>[1]</sup> For TMB301 Rollovers, BASELINE is the value recorded on Day 7 of the TMB-301 study. For TMB202 Rollovers, BASELINE is the value recorded on Day 0 of the TMB-202 study. Lab samples were not collected at the TMB-311 Screening for the Cohort 1 patients. EOS=End of Study visit conducted at Week 96.

 $\label{lem:westat} \begin{tabular}{ll} $\tt Created on DDMMYYYY) \\ {\tt S:\TMB311\DA\SAS\L\_LABOTH.SAS} \end{tabular}$ 

<sup>[2]</sup> L = Below lower limit of normal; H = Above upper limit of normal.

<sup>[3]</sup> Potentially Clinically Significant is defined as having a result either below the lower limit of normal or above the upper limit of normal.

# Listing 16.2.8.2 Viral Resistance Testing

Entry Inhibitors (Resistance)

| Treatment | Patient<br>ID | Visit | Visit<br>Date | Test Type | Reverse<br>Transcriptase<br>(Resistance) | Protease<br>(Resistance) | Integrase Genese<br>(Resistance) | Trop-<br>ism | Ibal-<br>izumab | Mara-<br>viroc | Enfu-<br>virt-<br>ide |
|---|---|---|---|---|---|---|---|---|---|---|---|
| C1:301/800mg | 311-xx- | xxx SCREEN | ING 2015-0 | 9-08 Geno | Abacavir (Y) Stavudine (P) Tenofovir (Y) Zidovudine (P) | Atazanavir (ATV) (N)<br>Tipranavir (P) | Dolutegravir (Y) | DM | Y | Y | Y |
| | | | | | Delavirdine (N) Didanosine (Y) Efavirenz (N) | Atazanavir (ATV/r) (P)<br>Darunavir (Y)<br>Fosamprenavir (P) | Elvitegravir (Y)<br>Raltegravir (Y) | | | | |
| | | | | Pheno | Abacavir (Y) Stavudine (Y) Tenofovir (Y) Zidovudine (Y) | Atazanavir (ATV) (Y)<br>Tipranavir (Y) | Dolutegravir (Y) | | | | |
| | | | | | Delavirdine (N) Didanosine (Y) Efavirenz (N) | Atazanavir (ATV/r) (Y)<br>Darunavir (Y)<br>Fosamprenavir (Y) | Elvitegravir (Y)<br>Raltegravir (Y) | | | | |
| | | WEEK 9 | 2015-11-03 | Geno | Abacavir (P)<br>Stavudine (N) | Atazanavir (ATV) (N)<br>Tipranavir (P) | Dolutegravir (Y) | DM | N | Y | Y |

(Continued)

Westat (Created on DDMMMYYYY) S:\TMB301\DA\SAS\L\_VRTEST.SAS

<sup>[1]</sup> EOS=End of Study visit conducted at Week 96.
[2] Note: Abbreviations for Resistance: Y = Sensitive, P = Partially Sensitive, N = Resistant

Listing 16.2.8.3 Vital Signs

| Treatment | Patient<br>ID | Visit | Visit<br>Date | Scheduled<br>Time Point | Time (hh:mm) | Height<br>(cm)<br>[2] | Weight<br>(kg)<br>[2] | Temp.<br>(C)<br>[2] | Rate<br>(bpm)<br>[2] | Resp. Rate (breaths/min) [2] | Systolic Blood<br>Pressure(mmHg)<br>[2] | Diastolic Blood<br>Pressure(mmHg)<br>[2] |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| C1:301/800mg | 311-XX-XXX | SCREENING | 2015-08-04 | | | 170 | 69 | 36.5 | 62 | 16 | 129 | 85 |
| | | DAY 0 | 2015-08-31 | | | | 69 | 36.9 | 81 | 16 | 108 | 68 |
| | | DAY 7 | 2015-09-08<br>2015-09-08 | | 10:45<br>12:00 | | | 36.9<br>36.8 | 74<br>76 | 15<br>16 | 127<br>110 | 76<br>69 |
| | | DAY 21 | 2015-09-22<br>2015-09-22 | | 10:00<br>11:05 | | | 36.9<br>36.8 | 82<br>80 | 15<br>15 | 103<br>115 | 68<br>72 |
| | | WEEK 5 | 2015-10-06<br>2015-10-06 | | 10:40<br>11:40 | | | 36.4*<br>36.8 | 67<br>76 | 16<br>15 | 126<br>122 | 83<br>72 |
| | | WEEK 7 | 2015-10-19<br>2015-10-19 | | 11:20<br>12:15 | | | 38.9*<br>37.1 | 117*<br>108 | 15<br>15 | 123<br>124 | 72<br>72 |
| | | WEEK 19 | 2016-01-14<br>2016-01-14 | | 12:45<br>13:25 | | | 36.8<br>36.7 | 79<br>78 | 16<br>16 | 108<br>109 | 65<br>70 |
| C1:202/800mg | 311-XX-XXX | SCREENING | 2015-08-05 | | | 179 | 83 | 36.6 | 69 | 15 | 124 | 85 |

<sup>[1]</sup>EOS=End of Study visit conducted at Week 96.

Westat (Created on DDMMMYYYY)
S:\TMB301\DA\SAS\L VITALS.SAS

<sup>[2]\*</sup>Denotes Potentially Clinically Significant Vital Signs outside of these ranges: Temperature: 36.44-37.22 C; Pulse: 60-110 BPM; Respiration rate: 12-20 breaths per minute; Blood Pressure: Systolic 100-140 mmHg; Diastolic 60-90 mmHg

Listing 16.2.8.4 Physical Examinations

| Treatment | Patient<br>ID | Visit | Visit Date | Performed<br>at Visit | Body System [1] | Status (Details) |
|---|---|---|---|---|---|---|
| Treatment | 15 | VISIC | VISIC Date | at visit | Body System [1] | Status (Details) |
| C1:301/800mg | 311-XX-XXX | Screening | DDMONYYYY | Yes/No | HEENT | Normal/Abnormal/Not Done |
| | | | | | Cardiovascular | xxx |
| | | | | | Musculoskeletal | xxx |
| | | | | | Lymphatic | xxx |
| | | | | | Respiratory | xxx |
| | | | | | Gastrointestinal | xxx |
| | | | | | Skin | xxx |

Neurological

Additional PE Findings

| C1:202/800mg | 311-xx-xxx | Day 0 | DDMONYYYY | Yes/No | Cardiovascular | Normal/Abnormal/Not Done |
|---|---|---|---|---|---|---|
| | | | | | Lymphatic | xxx |
| | | | | | Respiratory | xxx |
| | | | | | Abdomen | xxx |
| | | | | | Extremities | xxx |
| | | | | | Neurological | xxx |
| | | | | | Additional PE Findings | xxx |

<sup>[1]</sup>A complete physical examination is performed only at <list correct visits>. An abbreviated physical examination is performed at other visits.

Westat (Created on DDMMYYYY)
S:\TMB311\DA\SAS\L\_PHYSEXAM.SAS

Listing 16.2.9
Extent of Treatment Exposure

| Treatment | Patient<br>ID | Start Date of<br>Ibalizumab | Last Date of<br>Ibalizumab* | Years on<br>Ibalizumab |
|---|---|---|---|---|
| C1:301/800mg | 311-XX-XXX | 04MAR2016 | 21FEB2017 | 1.0 |
| C1:202/800mg | 311-XX-XXX | 23MAR2016 | 23FEB2017 | 0.9 |
| C1:202/2000mg | 311-XX-XXX | 16JUN2015 | 10FEB2017 | 1.7 |
| C2:800mg | 311-XX-XXX | 19AUG2015 | 15FEB2017 | 1.5 |

<sup>\*</sup>Last Dose recorded prior to the Data Cutoff Date.

Westat (Created on DDMMMYYYY) S:\TMB311\DA\SAS\L\_TRTEXP.SAS